CLINICAL TRIAL: NCT02655237
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-385 40 mg Compared With Leuprorelin in the Treatment of Uterine Fibroids
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Relugolix (TAK-385) 40 mg Compared With Leuprorelin in the Treatment of Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-385/CCT-002; U1111-1178-0989 (Registry Identifier: WHO); JapicCTI-163128 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Uterine Fibroids
Keywords: Drug Therapy
MeSH Terms: conditions — Leiomyoma | interventions — relugolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relugolix 40 mg (Experimental): Relugolix placebo matching tablets, orally, once daily along with leuprorelin acetate placebo matching injection, SC, once in 4 weeks for 3 to 6 weeks in run-in period followed by relugolix 40 mg, tablets, orally, once daily and leuprorelin acetate placebo matching injection, SC, once in 4 weeks for 24 weeks in treatment period.
  Interventions: Drug: Relugolix; Drug: Relugolix Placebo; Drug: Leuprorelin Placebo
- Leuprorelin 1.88 mg or 3.75 mg (Active Comparator): Relugolix placebo matching tablets, orally, once daily along with leuprorelin acetate placebo matching injection, SC, once in 4 weeks for 3 to 6 weeks in run-in period followed by leuprorelin acetate 1.88 mg or 3.75 mg, injection, SC, once in 4 weeks and relugolix placebo matching tablets, orally, once daily for 24 weeks in treatment period.
  Interventions: Drug: Relugolix Placebo; Drug: Leuprorelin; Drug: Leuprorelin Placebo

INTERVENTIONS:
Drug: Relugolix — Relugolix tablets
  Other Names: TAK-385
  Arms: Relugolix 40 mg
Drug: Relugolix Placebo — Relugolix placebo-matching tablets
Drug: Leuprorelin — Leuprorelin injection
  Arms: Leuprorelin 1.88 mg or 3.75 mg
Drug: Leuprorelin Placebo — Leuprorelin placebo-matching injections

SUMMARY:
The purpose of this study is to evaluate the efficacy of Relugolix (TAK-385) 40 mg administered orally once daily for 12 weeks, compared with leuprorelin injection (once every 4 weeks, 1.88 mg or 3.75 mg subcutaneously [SC]/time) in patients with uterine fibroids.

DETAILED DESCRIPTION:
The drug tested in this study was called Relugolix (TAK-385). Relugolix was tested to treat people who had uterine fibroids.

The study enrolled 281 patients. Participants received relugolix placebo and leuprorelin acetate placebo in run in period for 3 to 6 weeks. After run-in period, participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in 1:1 ratio:

* Relugolix 40 mg
* Leuprorelin 1.88 or 3.75 mg

Participants received relugolix tablets once daily along with leuprorelin 1.88 mg or 3.75 mg subcutaneous injection once in 4 weeks for 24 weeks in treatment period.

This multi-center trial was conducted in Japan. The overall time to participate in this study was approximately 32 to 40 weeks including run-in period of 3 to 6 weeks and a treatment period of 24 weeks. Participants will make multiple visits to the clinic, and a final visit 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Entering the Screening (at VISIT 1)

1. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. Prior to VISIT 1, the participant has a diagnosis of uterine fibroids confirmed by transvaginal ultrasound, abdominal ultrasound, magnetic resonance imaging (MRI), computed tomography (CT), or laparoscopy, and has never received any surgical treatment for the myoma (measurable noncalcified myoma with the longest diameter of ≥ 3 cm).
4. The participant is a premenopausal Japanese woman.
5. The participant is aged 20 years or older on the day of signing and dating the informed consent form.
6. The participant has 1 or more measurable noncalcified myomas with the longest diameter of ≥ 3 cm confirmed by transvaginal ultrasound.
7. The participant has experienced 1 or more regular menstrual cycles (25 to 38 days) immediately prior to VISIT 1 and that should include menstrual bleeding for at least 3 consecutive days.
8. The participant who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the study.

   Inclusion Criteria for Entering the Run-in (at VISIT 2)
9. The participant has experienced regular menstrual cycles (25 to 38 days) immediately prior to VISIT 2 that should include menstrual bleeding of at least 3 consecutive days (at least 2 regular menstruation cycles to be confirmed by Inclusion criteria #7 and #9).

   Inclusion Criteria for Entering the Treatment (at VISIT 3)
10. The participant has 1 or more measurable noncalcified myomas, with a longest diameter of ≥ 3 cm confirmed by transvaginal ultrasound (the same myoma should be measured as in Inclusion criterion #6).
11. The participant has a diagnosis of menorrhagia with a total Pictorial Blood loss Assessment Chart (PBAC) score of ≥ 120 in 1 menstrual cycle just before VISIT 3.
12. The participant has experienced regular menstrual cycles (25 to 38 days) after VISIT 1 that should include menstrual bleeding for at least 3 consecutive days (at least 3 regular menstruation cycles to be confirmed by Inclusion criteria #7, #9 and #12).

Exclusion Criteria:

1. The participant has received any investigational compound within 24 weeks prior to the start of the administration of the study medication for the Run-in (VISIT 2).
2. The participant has received relugolix (including placebo) in a previous clinical study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The participant has a previous or current history of blood disorders (eg, thalassemia, sickle cells anemia, folic-acid deficiency, and coagulopathy), excluding (latent) iron-deficiency anemia.
5. The participant has a known history of severe hypersensitivity or severe allergy to sanitary goods.
6. The participant has lower abdominal pain due to irritable bowel syndrome or severe interstitial cystitis.
7. The participant has a current history of thyroid gland disorder with irregular menstruation, or has a potential for irregular menstruation due to thyroid gland disorder, as determined by the investigator or subinvestigator.
8. The participant has a previous or current history of pelvic inflammatory disease within 8 weeks prior to VISIT 1.
9. The participant has a positive Pap smear test result obtained within 1 year prior to VISIT 1 (if there are no previous test results, those who were judged positive in the test conducted before VISIT 2).
10. The participant has a history of panhysterectomy or bilateral oophorectomy.
11. The participant has had markedly abnormal uterine bleeding or anovulatory bleeding, as determined by the investigator or subinvestigator.
12. The participant has a malignant tumor or a history of a malignant tumor within 5 years prior to VISIT 1.
13. The participant has been treated with any of the following drugs (excluding drugs for external use and dietary supplements) within 4 weeks prior to VISIT 2: anti-coagulant drugs, anti-platelet drugs, tranexamic acid, selective estrogen receptor modulators (SERMs), activated vitamin D preparations, other vitamin D preparations, calcitonin, ipriflavone, steroid hormones, vitamin K preparations, teriparatide, or denosumab.
14. The participant has been treated with any of the following drugs within 8 weeks prior to VISIT 2: oral contraceptive or sex hormone preparations (norethindrone, norethisterone, medroxyprogesterone, estrogen, or other progestins), and within 16 weeks prior to VISIT 2: gonadotropin-releasing hormone (GnRH) analogues, dienogest, danazol, or aromatase inhibitors (for 1- and 3-month sustained-release preparations, within 20 and 28 weeks prior to VISIT 2, respectively).
15. The participant has been treated with a bisphosphonate preparation within 24 weeks prior to VISIT 2.
16. The participant has a previous or current history of hypersensitivity or allergies to leuprorelin, synthetic GnRH, GnRH agonists or GnRH antagonists, or has a previous or current history of severe hypersensitivity or severe allergy to other drugs.
17. The participant has nondiagnosable abnormal genital bleeding.
18. Female participant who is pregnant, lactating, or intending to become pregnant or to donate ova prior to the signing of informed consent, during the study period, or within 1 month after the end of the study.
19. The participant has a previous or current history of osteoporosis, osteopenia, or other metabolic bone diseases.
20. The participant has clinically significant cardiovascular disease (eg, myocardial infarction or unstable angina pectoris within 24 weeks prior to VISIT 1) or uncontrollable hypertension (eg, resting systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg at Screening and Run-in).
21. The participant is inappropriate for participation in this study based on standard 12-lead electrocardiogram (ECG) findings, as determined by the investigator or subinvestigator.
22. The participant has active liver disease or jaundice, or with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin (total bilirubin) > 1.5 times the upper limit of normal (ULN) in the clinical laboratory tests at VISITs 1 and 2.
23. The participant has previous or current history of diseases considered to be inappropriate for participation in this study, including severe hepatic impairment, jaundice, renal impairment, cardiovascular disease, endocrine system disease, metabolic disorder, pulmonary disease, gastrointestinal disease, neurological disease, urological disease, immune disease, or mental disorder (especially depression-like symptoms) or suicide attempt resulting from a mental disorder.
24. The participant has a previous or current history of drug abuse (defined as any illicit drug use) or alcohol abuse.
25. The participant is inappropriate for participation in this study for other reasons, as determined by the investigator or subinvestigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (25):
- Japan (25):
  - Nagoya, Aichi-ken
  - Matsudo, Chiba
  - Kouriyama, Fukushima
  - Ebetsu, Hokkaido
  - Sapporo, Hokkaido
  - Kako-gun, Hyōgo
  - Nishinomiya, Hyōgo
  - Kawasaki, Kanagawa
  - Yamato, Kanagawa
  - Yokohama, Kanagawa
  - Ibaraki, Osaka
  - Sakai, Osaka
  - Suita, Osaka
  - Yao, Osaka
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuou-ku, Tokyo
  - Minato-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Suginami-ku, Tokyo
  - Taitou-ku, Tokyo
  - Kagoshima
  - Kyoto
  - Osaka
  - Saitama

REFERENCES:
- [Derived] Osuga Y, Enya K, Kudou K, Tanimoto M, Hoshiai H. Oral Gonadotropin-Releasing Hormone Antagonist Relugolix Compared With Leuprorelin Injections for Uterine Leiomyomas: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):423-433. doi: 10.1097/AOG.0000000000003141. PMID 30741797

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 34 investigative sites in Japan from 05 March 2016 to 25 September 2017.
Pre-assignment Details: Participants with a diagnosis of uterine fibroids were enrolled in 1 of 2 (Relugolix once daily and Leuprorelin once in 4 weeks) treatment groups.
Groups:
- Relugolix 40 mg: Relugolix placebo matching tablets, orally, once daily along with leuprorelin acetate placebo matching injection, subcutaneously (SC), once in 4 weeks for 3 to 6 weeks in run-in period followed by relugolix 40 mg, tablets, orally, once daily and leuprorelin acetate placebo matching injection, SC, once in 4 weeks for 24 weeks in treatment period.
- Leuprorelin 1.88 mg or 3.75 mg: Relugolix placebo matching tablets, orally, once daily along with leuprorelin acetate placebo matching injection, subcutaneously (SC), once in 4 weeks for 3 to 6 weeks in run-in period followed by leuprorelin acetate 1.88 mg or 3.75 mg, injection, SC, once in 4 weeks and relugolix placebo matching tablets, orally, once daily for 24 weeks in treatment period.
Period: Overall Study
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Started | 139 | 142
Completed | 122 | 131
Not Completed | 17 | 11
Not completed — Adverse Event | 10 | 7
Not completed — Protocol Deviation | 2 | 0
Not completed — Withdrawal by Participant | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Recovery Leading to Surgery | 2 | 1
Not completed — Reduction of Hemoglobin Concentration | 1 | 0
Not completed — Randomized but Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg | Total
Number analyzed (Participants) | 139 | 142 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (4.98) | 42.6 (5.27) | 42.9 (5.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 142 | 281
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 139 | 142 | 281
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 159.8 (5.29) | 159.4 (5.23) | 159.6 (5.25)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  kilogram (kg)
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 58.16 (9.167) | 59.53 (9.907) | 58.85 (9.557)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2] Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  kilogram per square meter (kg/m^2)
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 22.78 (3.506) | 23.43 (3.657) | 23.11 (3.592)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 96 | 89 | 185
  Current Smoker | 19 | 26 | 45
  Ex-Smoker | 24 | 27 | 51
Birth Experience [Count of Participants; unit: Participants]
  Had Birth Experience | 74 | 75 | 149
  Had No Birth Experience | 65 | 67 | 132
Type of Uterine Fibroid [Count of Participants; unit: Participants]
  Subserosal Fibroid | 54 | 53 | 107
  Intramural Fibroid | 117 | 112 | 229
  Submucosal Fibroid | 13 | 20 | 33
Stopped Any Medications for Uterine Fibroids [Count of Participants; unit: Participants]
  Had Stopped Any Medications | 30 | 37 | 67
  Had Not Stopped Any Medications | 109 | 105 | 214
Any Surgery for Uterine Fibroids [Count of Participants; unit: Participants]
  Had Any Surgery for Uterine Fibroids | 18 | 11 | 29
  Had Not Any Surgery for Uterine Fibroids | 121 | 131 | 252
Volume of Myoma [Mean (Standard Deviation); unit: cm^3] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  cm^3
    number analyzed (Participants) | 137 | 142 | 279
    (all) | 117.41 (126.533) | 122.25 (124.270) | 119.87 (125.184)
Volume of Uterus [Mean (Standard Deviation); unit: cm^3] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  cm^3
    number analyzed (Participants) | 136 | 139 | 275
    (all) | 406.25 (392.354) | 379.07 (331.568) | 392.51 (362.495)
Pictorial Blood Loss Assessment Chart (PBAC) Score [Mean (Standard Deviation); unit: score on a scale] — PBAC score was used to measure volume of menstrual blood loss. Participants used sanitary products designated by sponsor and recorded numbers of tampons or towels used, clots and flooding in patient diary. Three diagrams used which represented a lightly, moderately stained or completely saturated pad/tampon. Following scores assigned: 1) 1, 5, or 20 points for each pad; 2) 1, 5, or 10 points for each tampon; 3) 1 or 5 points for each blood clot of <1 cm/=1 cm/>1 in longest diameter; 4) 5 points for each episode of flooding. The total PBAC score (sum of points) ranges from 0 to >500. Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  score on a scale
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 254.3 (155.28) | 263.7 (171.33) | 259.1 (163.39)
Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: score on a scale] — Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain. Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  score on a scale
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 0.63 (0.790) | 0.56 (0.559) | 0.59 (0.682)
Uterine Fibroid Symptom and Quality of Life (UFS-QOL) Score: Symptom Severity [Mean (Standard Deviation); unit: score on scale] — UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total symptom severity score is ranging from 0 to 100. The higher scores indicate greater severity. Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  score on scale
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 28.4 (14.38) | 29.7 (15.18) | 29.1 (14.78)
UFS-QOL Score: Health Related Quality of Life (HRQL) Total [Mean (Standard Deviation); unit: score on a scale] — UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total HRQL score is ranging from 0 to 100. The higher scores indicate better QOL. Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  score on a scale
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 80.2 (16.73) | 76.8 (19.57) | 78.5 (18.27)
Hemoglobin [Mean (Standard Deviation); unit: Gram per deciliter (g/dL)] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  Gram per deciliter (g/dL)
    number analyzed (Participants) | 138 | 142 | 280
    (all) | 11.49 (1.368) | 11.62 (1.377) | 11.56 (1.372)
Dosage of Leuprorelin Vial [Count of Participants; unit: Participants] — Population: Here, number analyzed indicates participants who were evaluated for this baseline characteristic.
  Participants
    1.88 mg: number analyzed (Participants) | 138 | 142 | 280
    1.88 mg | 121 | 124 | 245
    3.75 mg: number analyzed (Participants) | 138 | 142 | 280
    3.75 mg | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total PBAC Score of <10 From Week 6 to 12
Description: PBAC score was used to measure volume of menstrual blood loss. Participants used sanitary products designated by sponsor and recorded the numbers of tampons or towels used, clots and flooding in patient diary. Three diagrams used which represented a lightly, moderately stained or completely saturated pad/tampon. Following scores assigned: 1) 1, 5, or 20 points for each pad; 2) 1, 5, or 10 points for each tampon; 3) 1 or 5 points for each blood clot of <1 cm/=1 cm/>1 in longest diameter; 4) 5 points for each episode of flooding. The total PBAC score (sum of points) ranges from 0 to >500.
Time Frame: Week 6 to 12
Population: Full analysis set (FAS) included all participants who were randomized and received at least 1 dose of the study drug for the treatment period. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
percentage of participants | 82.2 [75.773 to 88.672] | 83.1 [76.935 to 89.263]
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Test type: Non-Inferiority — The point estimate and 2-sided 95% confidence interval of the difference in the percentage were calculated between Relugolix 40 mg group and leuprorelin group (Relugolix 40 mg group - leuprorelin group), using Farrington and Manning (FM) method. If the lower boundary of the 95% CI was greater or equal to the non-inferiority margin of -15%, then the non-inferiority of Relugolix 40 mg to leuprorelin was concluded; p = 0.0013, Farrington and Manning (FM); Difference in percentage = -0.9, 95% CI 2-sided [-10.098 to 8.346] — Relugolix 40 mg-Leuprorelin

2. Secondary Outcome: Percentage of Participants With Total PBAC Score of <10 From Week 2 to 6
Description: as for outcome 1
Time Frame: Week 2 to 6
Population: FAS included all participants who were randomized and received at least 1 dose of the study drug for the treatment period. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
percentage of participants | 64.2 | 31.7
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Test type: Other — The point estimate and 2-sided 95% confidence interval of the difference in the percentage were calculated between relugolix 40 mg group and leuprorelin group, using FM method with the non-inferiority margin of -15%. The confidence interval was presented in a descriptive manner and not for the purpose of statistical inference; Difference in percentage = 32.5, 95% CI 2-sided [20.953 to 44.134] — Relugolix 40 mg-Leuprorelin

3. Secondary Outcome: Percentage of Participants With Total PBAC Score of <10 From Week 18 to 24
Description: as for outcome 1
Time Frame: Week 18 to 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
percentage of participants | 84.1 | 94.7
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; Difference in percentage = -10.6, 95% CI 2-sided [-18.337 to -2.883] — Relugolix 40 mg-Leuprorelin

4. Secondary Outcome: Percentage of Participants With Total PBAC Score of <10 for 6 Weeks Before the Final Dose of Study Drug
Description: as for outcome 1
Time Frame: For 6 weeks before the final dose of study drug (up to Week 24)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
percentage of participants | 79.0 | 92.3
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; Difference in percentage = -13.3, 95% CI 2-sided [-21.418 to -5.118] — Relugolix 40 mg-Leuprorelin

5. Secondary Outcome: Percent Change From Baseline in Myoma Volumes at Weeks 2, 4, 8, 12 and 24
Description: A transvaginal ultrasound was performed to determine myoma volumes. Only the largest myoma among those measurable at visit 1 was measured throughout the study. On the assumption that the myoma was spheroids, the myoma volumes were calculated using 3 diameters (D1, D2, and D3). D1: the longest diameter of the myoma; D2: the longest diameter of the myoma which was perpendicular to D1; D3: the diameter of the myoma which crossed the intersection of D1 and D2 (intersection "Z") and was perpendicular to D1/D2 plane. The formula used for calculation is Myoma volume= D1*D2*D3*π/6.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
cm^3
  Change at Week 2: number analyzed (Participants) | 135 | 142
  Change at Week 2 | -18.74 (31.849) | -6.68 (33.377)
  Change at Week 4: number analyzed (Participants) | 136 | 142
  Change at Week 4 | -24.99 (46.374) | -22.44 (31.935)
  Change at Week 8: number analyzed (Participants) | 132 | 141
  Change at Week 8 | -35.92 (39.546) | -40.62 (25.036)
  Change at Week 12: number analyzed (Participants) | 128 | 140
  Change at Week 12 | -43.28 (33.849) | -46.87 (24.067)
  Change at Week 24: number analyzed (Participants) | 124 | 132
  Change at Week 24 | -49.75 (34.331) | -53.71 (24.257)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 2; Test type: Other — The mean differences in the percent changes from baseline between relugolix 40 mg and leuprorelin group and the two-sided 95% confidence intervals were calculated; Mean Difference (Each Visit) = -12.05, 95% CI 2-sided [-19.778 to -4.330] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 4; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = -2.55, 95% CI 2-sided [-11.916 to 6.819] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 8; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = 4.69, 95% CI 2-sided [-3.141 to 12.529] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 12; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = 3.59, 95% CI 2-sided [-3.433 to 10.605] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 5: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 24; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = 3.96, 95% CI 2-sided [-3.319 to 11.245] — Relugolix 40 mg-Leuprorelin

6. Secondary Outcome: Percent Change From Baseline in Uterine Volumes at Weeks 2, 4, 8, 12 and 24
Description: A transvaginal ultrasound was performed for determination of uterine volumes. On the assumption that the uterus was spheroids, the uterine volumes were calculated using 3 diameters (D1, D2, and D3) measured as shown below: D1: the longest diameter of the uterus (unit of length: cm); D2: the longest diameter of the uterus which was perpendicular to D1 (unit of length: cm); D3: the diameter of the uterus which crossed the intersection of D1 and D2 (intersection "Z") and was perpendicular to D1/D2 plane (unit of length: cm). The formula used for calculation is Uterine volume=D1*D2*D3*π/6.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
cm^3
  Change at Week 2: number analyzed (Participants) | 133 | 138
  Change at Week 2 | -22.05 (17.870) | -6.90 (27.984)
  Change at Week 4: number analyzed (Participants) | 135 | 139
  Change at Week 4 | -28.07 (23.965) | -17.80 (34.058)
  Change at Week 8: number analyzed (Participants) | 131 | 138
  Change at Week 8 | -34.73 (22.507) | -33.83 (27.882)
  Change at Week 12: number analyzed (Participants) | 127 | 137
  Change at Week 12 | -39.79 (24.454) | -38.85 (25.157)
  Change at Week 24: number analyzed (Participants) | 123 | 129
  Change at Week 24 | -44.87 (29.214) | -45.73 (27.778)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 2; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = -15.15, 95% CI 2-sided [-20.786 to -9.509] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 4; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = -10.27, 95% CI 2-sided [-17.291 to -3.246] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 8; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = -0.89, 95% CI 2-sided [-6.996 to 5.209] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 12; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = -0.94, 95% CI 2-sided [-6.964 to 5.076] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 5: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 24; Test type: Other — [test comment as in outcome 5, analysis 1]; Mean Difference (Each Visit) = 0.86, 95% CI 2-sided [-6.206 to 7.935] — Relugolix 40 mg-Leuprorelin

7. Secondary Outcome: Change From Baseline in Hemoglobin at Weeks 4, 8, 12, 16, 20, 24 and Follow up
Description: Anemia-related measurements consisted of hemoglobin, which were determined at the central laboratory.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24 and Follow up (up to Week 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
g/dL
  Change at Week 4: number analyzed (Participants) | 137 | 142
  Change at Week 4 | 0.79 (0.763) | 0.60 (0.789)
  Change at Week 8: number analyzed (Participants) | 133 | 141
  Change at Week 8 | 1.20 (1.043) | 1.10 (0.925)
  Change at Week 12: number analyzed (Participants) | 129 | 140
  Change at Week 12 | 1.38 (1.134) | 1.31 (1.000)
  Change at Week 16: number analyzed (Participants) | 129 | 136
  Change at Week 16 | 1.40 (1.190) | 1.42 (0.978)
  Change at Week 20: number analyzed (Participants) | 125 | 132
  Change at Week 20 | 1.47 (1.264) | 1.58 (1.033)
  Change at Week 24: number analyzed (Participants) | 122 | 131
  Change at Week 24 | 1.56 (1.281) | 1.65 (1.116)
  Change at Follow-Up (up to Week 28): number analyzed (Participants) | 136 | 141
  Change at Follow-Up (up to Week 28) | 1.25 (1.301) | 1.75 (1.182)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 4; Test type: Other — The mean differences in the change from baseline between relugolix 40 mg and leuprorelin groups and the two-sided 95% confidence intervals were calculated for each visit; Mean Difference (Each Visit) = 0.20, 95% CI 2-sided [0.015 to 0.381] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 8; Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = 0.10, 95% CI 2-sided [-0.135 to 0.333] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 12; Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = 0.07, 95% CI 2-sided [-0.189 to 0.323] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 16; Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = -0.01, 95% CI 2-sided [-0.275 to 0.251] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 5: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 20; Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = -0.10, 95% CI 2-sided [-0.386 to 0.180] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 6: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 24; Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = -0.09, 95% CI 2-sided [-0.385 to 0.209] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 7: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Follow up (up to Week 28); Test type: Other — [test comment as in outcome 7, analysis 1]; Mean Difference (Each Visit) = -0.49, 95% CI 2-sided [-0.787 to -0.199] — Relugolix 40 mg-Leuprorelin

8. Secondary Outcome: Numerical Rating Scale (NRS) Score
Description: Pain symptoms were evaluated using the NRS score. NRS score is a self-reported instrument assessing pain from 0 to 10. Higher scores reflect greater level of pain.
Time Frame: From Week 6 to 12, from Week 2 to 6, from Week 18 to 24, and for 6 weeks before the final dose (up to Week 24)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
score on a scale
  Week 6 to 12: number analyzed (Participants) | 135 | 142
  Week 6 to 12 | 0.21 (0.500) | 0.14 (0.363)
  Week 2 to 6: number analyzed (Participants) | 137 | 142
  Week 2 to 6 | 0.32 (0.707) | 0.27 (0.489)
  Week 18 to 24: number analyzed (Participants) | 126 | 133
  Week 18 to 24 | 0.12 (0.308) | 0.11 (0.289)
  For 6 weeks before the final dose (up to Week 24) | 0.14 (0.359) | 0.12 (0.327)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 6 to 12; Test type: Other — Two-sided 95% confidence interval of the difference was calculated between relugolix 40 mg and leuprorelin group; Mean Difference (Each Visit) = 0.07, 95% CI 2-sided [-0.032 to 0.174] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 2 to 6; Test type: Other — Two-sided 95% confidence interval of the difference was calculated between relugolix 40 mg and leuprorelin group; Mean Difference (Each Visit) = 0.05, 95% CI 2-sided [-0.089 to 0.197] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 18 to 24; Test type: Other — Two-sided 95% confidence interval of the difference was calculated between relugolix 40 mg and leuprorelin group; Mean Difference (Each Visit) = 0.01, 95% CI 2-sided [-0.060 to 0.086] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; For 6 Weeks Before the Final Dose (up to Week 24); Test type: Other — Two-sided 95% confidence interval of the difference was calculated between relugolix 40 mg and leuprorelin group; Mean Difference (Each Visit) = 0.02, 95% CI 2-sided [-0.063 to 0.099] — Relugolix 40 mg-Leuprorelin

9. Secondary Outcome: Change From Baseline in Uterine Fibroid Symptom and Quality of Life (UFS-QOL)- Symptom Severity Score at Weeks 4, 8, 12, 16, 20, 24 and Follow-up
Description: UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total symptom severity score is ranging from 0 to 100. The higher scores indicate greater severity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24 and Follow-up (up to Week 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
score on a scale
  Change at Week 4: number analyzed (Participants) | 137 | 142
  Change at Week 4 | -5.5 (14.11) | -4.5 (16.09)
  Change at Week 8: number analyzed (Participants) | 133 | 141
  Change at Week 8 | -19.5 (14.47) | -17.2 (16.91)
  Change at Week 12: number analyzed (Participants) | 129 | 140
  Change at Week 12 | -21.0 (14.93) | -23.0 (14.66)
  Change at Week 16: number analyzed (Participants) | 129 | 136
  Change at Week 16 | -21.4 (14.76) | -24.4 (14.04)
  Change at Week 20: number analyzed (Participants) | 125 | 132
  Change at Week 20 | -21.9 (14.97) | -24.3 (14.87)
  Change at Week 24: number analyzed (Participants) | 122 | 131
  Change at Week 24 | -22.5 (15.17) | -25.3 (14.52)
  Change at Follow-Up (up to Week 28): number analyzed (Participants) | 136 | 141
  Change at Follow-Up (up to Week 28) | -20.6 (16.83) | -25.4 (14.04)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 4; Test type: Other — The mean differences in the observed values between relugolix 40 mg and leuprorelin group and the two-sided 95% confidence intervals were calculated for each visit; Mean Difference (Each Visit) = -2.5, 95% CI 2-sided [-6.39 to 1.43] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 8; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = -4.0, 95% CI 2-sided [-6.68 to -1.31] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 12; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.2, 95% CI 2-sided [-1.99 to 2.36] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 16; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 1.3, 95% CI 2-sided [-0.68 to 3.28] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 5: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 20; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.3, 95% CI 2-sided [-1.80 to 2.32] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 6: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 24; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.5, 95% CI 2-sided [-1.48 to 2.52] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 7: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Follow-Up (up to Week 28); Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 3.4, 95% CI 2-sided [1.08 to 5.77] — Relugolix 40 mg-Leuprorelin

10. Secondary Outcome: Change From Baseline in Uterine Fibroid Symptom and Quality of Life (UFS-QOL)- HRQL Total Scores at Weeks 4, 8, 12, 16, 20, 24 and Follow-up
Description: UFS-QOL was a 37-item self-reporting tool for evaluating QOL in participants with uterine fibroid. It includes eight symptom-related questions and 29 HRQL questions across six subscales (concern, activities, energy/mood, control, self-consciousness, sexual function). The total HRQL score is ranging from 0 to 100. The higher scores indicate better QOL.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24 and Follow-up (up to Week 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
score on a scale
  Change at Week 4: number analyzed (Participants) | 137 | 142
  Change at Week 4 | 2.4 (12.42) | 3.5 (12.89)
  Change at Week 8: number analyzed (Participants) | 133 | 141
  Change at Week 8 | 8.1 (14.48) | 9.5 (16.78)
  Change at Week 12: number analyzed (Participants) | 129 | 140
  Change at Week 12 | 10.4 (15.01) | 13.3 (17.99)
  Change at Week 16: number analyzed (Participants) | 129 | 136
  Change at Week 16 | 10.9 (14.43) | 14.3 (18.31)
  Change at Week 20: number analyzed (Participants) | 125 | 132
  Change at Week 20 | 11.5 (14.65) | 14.5 (17.59)
  Change at Week 24: number analyzed (Participants) | 122 | 131
  Change at Week 24 | 12.0 (14.91) | 15.8 (18.13)
  Change at Follow-Up (up to Week 28): number analyzed (Participants) | 136 | 141
  Change at Follow-Up (up to Week 28) | 10.9 (16.53) | 15.7 (18.08)
Statistical Analysis 1: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 4; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 2.3, 95% CI 2-sided [-1.66 to 6.34] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 2: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 8; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 2.7, 95% CI 2-sided [-0.37 to 5.77] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 3: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 12; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.9, 95% CI 2-sided [-1.84 to 3.61] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 4: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 16; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.1, 95% CI 2-sided [-2.61 to 2.79] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 5: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 20; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.8, 95% CI 2-sided [-1.74 to 3.41] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 6: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Week 24; Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = 0.3, 95% CI 2-sided [-2.07 to 2.71] — Relugolix 40 mg-Leuprorelin
Statistical Analysis 7: Comparison: Relugolix 40 mg vs Leuprorelin 1.88 mg or 3.75 mg; Follow-Up (up to Week 28); Test type: Other — [test comment as in outcome 9, analysis 1]; Mean Difference (Each Visit) = -1.4, 95% CI 2-sided [-3.96 to 1.09] — Relugolix 40 mg-Leuprorelin

11. Secondary Outcome: Number of Participants Who Had One or More Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants | 131 | 139

12. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Vital Signs
Description: Vital signs included sitting blood pressure (after the participant has rested for at least 5 minutes), body temperature (oral or tympanic measurement) (degree Celsius [°C]) and pulse (beats per minute [bpm]) is reported.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants
  Systolic Blood Pressure Lower (<85 mmHg) | 3 | 2
  Systolic Blood Pressure Upper (>180 mmHg) | 0 | 1
  Diastolic Blood Pressure Lower (<50 mmHg) | 5 | 5
  Diastolic Blood Pressure Upper (>110 mmHg) | 2 | 3
  Pulse Rate Lower (<50 bpm) | 0 | 1
  Body temperature Lower (<35.6 °C) | 23 | 23
  Body temperature Upper (>37.7 °C) | 1 | 0

13. Secondary Outcome: Number of Participants With TEAE Related to Weight
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to weight was reported.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With TEAE Related to Standard 12-Lead ECGs
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to ECG was reported.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Laboratory Test
Description: Number of participants with any markedly abnormal values in laboratory tests collected throughout study is reported. WBC = White blood cells, AST = Aspartate Aminotransferase, ALT = Alanine Aminotransferase, GGT = gamma-glutamyl transferase, ULN = upper limit of normal or upper reference limit.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants
  WBC Upper (>1.5×ULN×10^3 cells/μL) | 1 | 0
  Eosinophils Upper (>2×ULN×10^3 cells/μL) | 3 | 4
  Total cholesterol Upper (>300 mg/dL) | 6 | 4
  Triglycerides Upper (>2.5×ULN mg/dL) | 4 | 12
  Creatine kinase Upper (>5×ULN U/L) | 1 | 0
  AST Upper (>3×ULN U/L) | 2 | 0
  ALT Upper (>3×ULN U/L) | 3 | 2
  GGT Upper (>3×ULN U/L) | 10 | 6
  Hemoglobin A1c Upper (>7%) | 0 | 2

16. Secondary Outcome: Number of Participants With TEAE (Bone Density Decreased) Related to Bone Mineral Density
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to bone mineral density was reported.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants | 6 | 8

17. Secondary Outcome: Number of Participants With TEAE Related to Biochemical Bone Metabolism Markers
Description: Number of participants with TEAEs of which threshold was 5% or above in either treatment group related to biochemical bone metabolism markers was reported.
Time Frame: Up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
Number analyzed (Participants) | 138 | 142
Participants
  Bone Resorption Test Abnormal | 7 | 7
  Resorption Bone Increased | 7 | 8

ADVERSE EVENTS:
Time Frame: Up to Week 28
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Relugolix 40 mg | Leuprorelin 1.88 mg or 3.75 mg
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/138 | 2/142
Other Adverse Events (participants affected / at risk) | 123/138 | 134/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix 40 mg (N=138) | Leuprorelin 1.88 mg or 3.75 mg (N=142)
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix 40 mg (N=138) | Leuprorelin 1.88 mg or 3.75 mg (N=142)
Malaise (General disorders) | 8 | 5
Viral upper respiratory tract infection (Infections and infestations) | 39 | 46
Gamma-glutamyltransferase increased (Investigations) | 7 | 9
Bone density decreased (Investigations) | 6 | 8
Bone resorption test abnormal (Investigations) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 7 | 8
Headache (Nervous system disorders) | 21 | 14
Dizziness (Nervous system disorders) | 9 | 7
Somnolence (Nervous system disorders) | 7 | 6
Metrorrhagia (Reproductive system and breast disorders) | 68 | 93
Menorrhagia (Reproductive system and breast disorders) | 34 | 22
Genital haemorrhage (Reproductive system and breast disorders) | 7 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 | 15
Hot flush (Vascular disorders) | 59 | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT02655237/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02655237/SAP_001.pdf